CLINICAL TRIAL: NCT06504979
Title: Implementation of a Digital Tool for the Telematic Follow-up and Management of Emotional and Cognitive Sequelae Related to Post-intensive Care Syndrome: Impact on Quality of Life and Functionality
Brief Title: The Post Intensive Care Syndrome Follow-up and Management Study: the ICU Recovery Answers Project
Acronym: ICURA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Universitat de les Illes Balears (Other); Hospital Son Espases (Other); Fundació La Marató de TV3 (Other)
Responsible Party: Principal Investigator, Sol Fernandez-Gonzalo, Principal Investigator, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/3031
Record Dates: First submitted 2024-06-18; First posted 2024-07-17 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Post Intensive Care Syndrome; ICU Survivors; ICU Families
Keywords: Post-intensive Care Syndrome; ICU survivors; ICU families; Cognition; Emotional state
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICURA follow-up (Experimental)
  Interventions: Other: Telehealth follow-up of post-intensive care syndrome
- Standard Group (No Intervention)

INTERVENTIONS:
Other: Telehealth follow-up of post-intensive care syndrome — Using a telehealth platform for the detection of the emotional, neuropsychological and physical PICS-related sequelae along 12 months in ICU survivors
  Arms: ICURA follow-up

SUMMARY:
Critically ill survivors develop mental health, cognition, and mobility sequelae known as Post-Intensive Care Syndrome (PICS). Clinically significant symptoms of post-traumatic stress, depression, anxiety, and cognitive impairment are frequently observed at short- and long-term after ICU, impacting quality of life of the survivors and their relatives.

The main objective of the project is to optimize, implement and evaluate the impact in quality of life of a digital platform (ICURA) specifically designed for following-up and managing the mental health sequelae related to PICS in ICU survivors and their relatives during the one-year recovery phase.

Methods: Observational, prospective and multicenter study including two cohorts: 1) ICU patients' cohort (ICUcohort), and 2) ICU patients' family cohort (ICU-F-cohort). After ICU discharge, patients will be randomized to participate in a follow-up with ICURA vs. the standard follow-up.

Expected results: Critically ill survivors in the APPICS program after ICU will show better levels of functionality and quality of life than those participants in the usual follow-up. APPICS will contribute to enhancing the prognosis of emotional alterations during the 12 months after ICU both, in ICU survivors, and relatives. Analyzing risk factors, based on demographic and clinical data, will help to the early detection of long-term mental health difficulties in ICU survivors.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old) critically ill patients admitted to the ICU with or without need of invasive mechanical ventilation (IMV).

Exclusion Criteria:

* Non-authorization of the relatives and/or patient to inclusion in the study; neurocritical ICU patients.
* Severe neurological pathology (including dementia or focal brain damage with functional and cognitive impairment) prior to admission to the ICU.
* Severe psychiatric pathology (schizophrenia, bipolar disorder, major depressive disorder)
* Intellectual disability (IQ <80).
* Patients who develop secondary complications (infections, stroke, TBI or any non-transient acquired brain damage) after ICU discharge, that may compromise the results of the emotional and neuropsychological evaluation during the recovery phase
* Moderate-severe cognitive impairment (Short-IQCODE >85) that impair ICU patients an independent participation in the telematic follow up and accompaniment program
* Readmission to ICU within 12 months after discharge from ICU
* Idiomatic barrier (non spanish and/or catalan speaker)
* Patients with life expectancy <1 year or not subsidiaries of active treatment measures.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | 1 year
  12-Item Short Form Survey (SF-12) at 12 months after ICU discharge Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Functionality | 1 year
  WHO Short Disability Assessement Schedule (WHODAS 2.0) 12 months after ICU discharge. Scores range from 0 to 60, with higher scores indicating higher level of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut d'Investigació i Innovació Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: ICURA project website — https://www.tauli.cat/es/institut/projectes-i-xarxes/projectes-financats/icura/